CLINICAL TRIAL: NCT06938464
Title: The Preventive Effect of Probiotics in Pregnant Women With High-risk for Gestational Diabetes
Brief Title: Preventive Effect of Probiotics in GDM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Quzhou Maternal and Child Health Care Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-20230226-R
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Gestational Diabetes Mellitus (GDM)
MeSH Terms: conditions — Diabetes, Gestational | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The random number table is compiled by the investigator who is specially responsible for grouping and saved. The investigator packaged and coded drugs according to random number table, and recorded. The packaged and numbered drugs are stored in the enrollment office.
  When the participants meet the inclusion criteria by care providers (doctors), the enrollment office generates a random number for each subject. The participants received the package of drugs according to their random number, and the random number was recorded in the record book.
  If there are adverse events or the subjects request to withdraw from the trial, the investigator should uncover the blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Active Comparator): Probiotic powder 1 bag per day, as well as health guidance about diet and exercise. From recruitment until OGTT.
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Placebo 1 bag per day. Similar health guidance about diet and exercise. From recruitment until OGTT
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Probiotics powder including: Resistant dextrin, inulin, oligosaccharide, erythritol, Lactobacillus plantarum VB165, Bifidobacterium lactis VB301, Lactobacillus rhamnosus VB255, acerola cherry powder, citric acid
  Arms: Probiotics
Dietary Supplement: Placebo — placebo with similar appearance and smell but not containing probiotics
  Arms: Placebo

SUMMARY:
Gut microbiota is instrumental in the microbial and metabolic network of pregnant women, and is potentially related with gestational diabetes. Perinatal probiotic intervention contributes to improved glucose regulation during pregnancy. Our randomized, double-centered, placebo-controlled study is planned to recruit 334 pregnant women who is in high risk for gestational diabetes. They will be assumed randomly probiotic powder per day or placebo from 12-16th gestational weeks until Oral Glucose Tolerance Test (OGTT) at 24-28th gestational weeks. Perinatal outcomes about neonatal weight will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who meet the high-risk indicators for GDM and agree to participate in this study.

  1. included between 12-16 gestational weeks
  2. A woman was considered high risk when her pre-pregnancy BMI ≥ 24 kg/m^2, having family history of diabetes (type 1 or 2), GDM or PCOS (polycystic ovary syndrome) history, history of delivering macrosomia or stillbirth, or glucose in urine (+)

Exclusion Criteria:

1. Taking probiotics or prebiotics within the past month
2. Have a history of allergies to the drug components or similar drugs in this study
3. Having long-term smoking or drinking habits
4. Type 1 or type 2 diabetes patients with definite diagnosis before pregnancy
5. Diseases in other important organs such as heart, liver, and kidney
6. with clear digestive system diseases
7. Multiple pregnancy
8. with mental or cognitive impairments who are unable to complete this study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 334 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of gestational diabetes | 24-28th weeks gestation
  The number of cases and incidence of gestational diabetes according to OGTT

SECONDARY OUTCOMES:
The incidence of macrosomia | Delivery
  macrosomia refers to a newborn weighs more than 4 kg)
Weight gain during pregnancy (kg) | Delivery
  Weight gain during pregnancy (kg) = Maternal weight at delivery - weight pre-pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China